CLINICAL TRIAL: NCT04228419
Title: Study Evaluating Reverse Versus Anatomic Shoulder Arthroplasty Techniques in the Treatment of Osteoarthritis: Protocol
Brief Title: TSA vs RSA in Glenohumeral Osteoarthritis
Acronym: SERVASA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190674-01H
Record Dates: First submitted 2019-12-17; First posted 2020-01-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: arthroplasty; glenohumeral osteoarthritis; idiopathic osteoarthritis
MeSH Terms: interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Shoulder Arthroplasty (anatomic) (Active Comparator): TSA procedure involves replacing the worn-out ball and socket joint with prosthetic components.
  Interventions: Procedure: Total Shoulder Arthroplasty
- Reverse Shoulder Arthroplasty (Active Comparator): RSA procedure is similar to a TSA, however the orientation of the ball and socket joint is placed in the reverse position
  Interventions: Procedure: Reverse Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Total Shoulder Arthroplasty — Replacement of the shoulder joint (ball and socket, or humeral head and glenoid) using prosthetic components.
  Arms: Total Shoulder Arthroplasty (anatomic)
Procedure: Reverse Shoulder Arthroplasty — Replacement of the shoulder joint like the TSA, however the orientation of the ball and socket is reversed.
  Arms: Reverse Shoulder Arthroplasty

SUMMARY:
This study will compare total shoulder arthroplasty (TSA) reverse shoulder arthroplasty (RSA) procedures, in the context of a prospective, randomized-controlled trial to determine the optimal treatment in patients 65 years of age and older, and equal to or less than 15 degrees of glenoid retroversion, who have glenohumeral osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the shoulder is a disease resulting from the wearing down of cartilage over time. OA can be the cause of pain and dysfunction and is a growing occurrence in the investigator's aging population. TSA or RSA are common surgical procedures used to treat patients with shoulder OA. TSA is able to keep the "natural anatomy" of the shoulder and involves replacing the worn-out ball and socket shoulder joint with prosthetic components. TSA is performed today with high success rates, however, complication rates associated with TSA remain prevalent, particularly when the arthritis is associated with bone erosion on the glenoid (socket).

RSA is an alternative surgical procedure commonly used and involves replacing and reversing the ball and the socket (i.e. opposite of TSA). RSA is typically performed in patients with a rotator cuff deficiency and more severe OA. Though RSA procedures show marked increase in clinical and functional outcomes, evidence of its long-term results are sparse, and as such is typically reserved for when treating an older patient population.

Few research studies have compared these different surgical techniques to one another, in the older patient population.

This research will provide surgeons with new information regarding the best treatment for patients in this population.

This Randomized Controlled Trial (RCT) will compare TSA and RSA procedures in those 65 years of age and older, who have equal to or less than 15 degrees of glenoid retroversion, in an effort to determine which approach produces better functional outcomes and improved quality of life in this patient population.

Primary Objective: Determine the difference in disease specific quality of life between patients diagnosed with glenohumeral OA who undergo either a TSA or RSA as measured by the Western Osteoarthritis of the Shoulder (WOOS) score at 24-months and 5-years post-operative.

Secondary Objectives: i) Determine the difference in disease specific quality of life between patients diagnosed with a glenohumeral osteoarthritis who undergo a shoulder replacement with RSA or TSA as measured by the Constant score, the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES), the EuroQol Group EQ-5D-5L score, pain (using a Visual Analog Scale), and Subjective Shoulder Value (SSV) at 24-months and 5-years post-operative as well as adverse events, and health care utilization.

ii) To determine the survivorship of the components as measured by the degree of radiographic lucencies and component alignment determined by a CT scan at 1- and 5-years post-surgery.

Clinical Relevance: Shoulder OA results in pain and dysfunction, which negatively impacts quality of life. As such, determination of superior treatment approach will lead to significant improvement in quality of life, and cost savings through avoidance of recurrence and/or reoperation, as well as decreased morbidity for patients in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have failed standard non-surgical management of their idiopathic shoulder osteoarthritis who would benefit from a shoulder arthroplasty. Failed medical management will be defined as persistent pain and disability despite adequate standard non-operative management for 6 months. Medical management will be defined as:

   1. The use of drugs including analgesics and non-steroidal anti-inflammatory drugs
   2. Physiotherapy consisting of stretching, strengthening and local modalities (ultrasound, cryotherapy, etc.)
   3. Activity modification
2. Imaging, and intra-operative findings confirming advanced glenohumeral cartilage loss
3. Patients may present with a glenoid deficiency and </=15 degrees of retroversion
4. 65 years of age and older

Exclusion Criteria:

1. Active joint or systemic infection
2. Rotator cuff arthropathy
3. Significant muscle paralysis
4. Charcot's arthropathy
5. Major medical illness (life expectancy less than 1 year or unacceptably high operative risk)
6. Unable to understand the consent form/process
7. Pregnancy
8. Psychiatric illness that precludes informed consent
9. Unwilling to be followed for the duration of the study
10. Retroversion cannot be surgically corrected to within 10 degrees of neutral
11. History of previous shoulder surgery on affected side

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | 24-Months and 5-Years Post-Operative
  The Western Ontario Osteoarthritis of the Shoulder Index (WOOS) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WOOS is a patient-reported measure, 19-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.

SECONDARY OUTCOMES:
Standard CT Scans | 24-Months and 5-Years Post-Operative
  Radiological parameters will be examined using Computed Tomography (CT). These scans will be analyzed for abnormalities in component alignment, and evidence of lucencies or loosening. Higher incidence of loosening, or noted abnormalities will be compared between groups. A higher incidence indicates worse outcomes.
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES) | 24-Months and 5-Years Post-Operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Pain Level | 24-Months and 5-Years Post-Operative
  Subjective pain value of the shoulder will be assessed using a questionnaire. Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. The higher the score, the worse the outcome.
Subjective Shoulder Value | 24-Months and 5-Years Post-Operative
  A participant's subjective value on shoulder function will be assessed using a questionnaire. The overall functional value of the shoulder is written as a percentage from 0-100% of a normal shoulder. The higher the score, the better the outcome.
EuroQol EQ-5D-5L | 24-Months and 5-Years Post-Operative
  The EQ-5D-5L quality of life questionnaire is a brief, easy to administer generic health status questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (each question rated 1-5), lower scores indicate better outcome. It also includes a visual analogue scale for recording an individual's rating of their current health-related quality of life (scale 0 to 100), where a higher score indicates a better outcome.
Constant Score | 24-Months and 5-Years Post-Operative
  The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
Adverse Events (AE) and Serious Adverse Events (SAE) | 24-Months and 5-Years Post-Operative
  Rates of study adverse events or serious adverse events (e.g. number of reoperations) will be monitored and recorded and compared between study groups. A higher rate of adverse events indicates a worse outcome.
Health Care Utilization | 24-Months and 5-Years Post-Operative
  Health care utilization will be monitored and recorded using a questionnaire. These questions will include healthcare the patient accessed, cost of care, and medications taken during treatment. From this information, a cost-effectiveness analysis will be completed, which will adhere to the best practices for conducting and reporting of health economic evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital
Locations (4):
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Pan Am Clinic Foundation, Winnipeg, Manitoba
  - Kingston General Hospital (Site-Watkins 3), Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers, who are not participating in the study.